CLINICAL TRIAL: NCT04091490
Title: Dexamethasone, Cytarabine, Cisplatin and Nivolumab in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma (Nivo-DHAP-cHL)
Brief Title: Combination of Nivolumab and DHAP in Patients With Relapsed or Refractory Classical Hodgkin Lymphoma (Nivo-DHAP)
Acronym: Nivo-DHAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nivo-DHAP-cHL-1
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with relapsed/refractory Hodgkin's lymphoma (Experimental): A clinical study of safety and efficacy of treatment with Nivolumab and DHAP in patients with relapsed/refractory Hodgkin's lymphoma
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Combination of 2 cycles of Nivolumab as a monotherapy with 4 cycles of high-dose chemotherapy (DHAP chemoregimen) with Nivolumab
  Other Names: Opdivo

SUMMARY:
A clinical study of safety and efficacy of treatment with Nivolumab and DHAP in patients with relapsed/refractory Hodgkin's lymphoma

DETAILED DESCRIPTION:
A Clinical Study of Safety and Efficacy of Treatment With Nivolumab and Dexamethasone, Cytarabine and Cisplatin (DHAP) in Patients With Relapsed/Refractory Hodgkin's Lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically confirmed Hodgkin's lymphoma
* Measurable disease (at least one lesion that can be accurately measured in at least two dimensions with spiral CT scan, min > 15 mm in the longest diameter or > 10 mm in the short axis)
* World Health Organization (WHO) performance status < 2
* Relapsed or refractory to at least one prior treatment line
* No prior therapy with DHAP or Nivolumab
* No severe concurrent illness

Exclusion Criteria:

* History of HIV
* Active Hepatitis B or Hepatitis C infection
* Uncontrolled infection (requiring intravenous treatment) at the time of enrollment
* Pregnancy or breastfeeding
* Somatic or psychiatric disorder making the patient unable to sign informed consent
* Active or prior documented autoimmune disease requiring systemic treatment
* No receiving a live vaccine within 30 days prior to first dose of nivolumab
* History of non-infectious pneumonitis that required steroids
* Other malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) of Nivolumab and DHAP in patients with relapsed/refractory Hodgkin's lymphoma | up to 6 months
  Overall response rate (ORR), defined as proportion of patients with complete response (CR) or partial response (PR) in measurable lesions as defined by Lugano classification and duration of response

SECONDARY OUTCOMES:
Frequency of grade 3 or higher treatment-related adverse events by CTCAE 4.03 | up to 6 months
  Toxicity parameters based on NCI CTCAE 4.03 grades
Progression-Free Survival | up to 12 months
Overall Survival | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vladislav Sarzhevskiy, PhD, Principal Investigator — National Medical Surgical Center named after N. I. Pirogov of the Ministry of health of the Russian Federation
Locations (1):
- The Federal Budget-Funded Institution National Medical Surgical Center named after N. I. Pirogov of the Ministry of health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sasse S, Alram M, Muller H, Smardova L, Metzner B, Doehner H, Fischer T, Niederwieser DW, Schmitz N, Schafer-Eckart K, Raemaekers JM, Schmalz O, Tresckow BV, Engert A, Borchmann P. Prognostic relevance of DHAP dose-density in relapsed Hodgkin lymphoma: an analysis of the German Hodgkin-Study Group. Leuk Lymphoma. 2016 May;57(5):1067-73. doi: 10.3109/10428194.2015.1083561. Epub 2015 Dec 23. PMID 26693800
- [Background] Armand P, Engert A, Younes A, Fanale M, Santoro A, Zinzani PL, Timmerman JM, Collins GP, Ramchandren R, Cohen JB, De Boer JP, Kuruvilla J, Savage KJ, Trneny M, Shipp MA, Kato K, Sumbul A, Farsaci B, Ansell SM. Nivolumab for Relapsed/Refractory Classic Hodgkin Lymphoma After Failure of Autologous Hematopoietic Cell Transplantation: Extended Follow-Up of the Multicohort Single-Arm Phase II CheckMate 205 Trial. J Clin Oncol. 2018 May 10;36(14):1428-1439. doi: 10.1200/JCO.2017.76.0793. Epub 2018 Mar 27. PMID 29584546
- [Result] Josting A, Rudolph C, Reiser M, Mapara M, Sieber M, Kirchner HH, Dorken B, Hossfeld DK, Diehl V, Engert A; Participating Centers. Time-intensified dexamethasone/cisplatin/cytarabine: an effective salvage therapy with low toxicity in patients with relapsed and refractory Hodgkin's disease. Ann Oncol. 2002 Oct;13(10):1628-35. doi: 10.1093/annonc/mdf221. PMID 12377653